CLINICAL TRIAL: NCT02555722
Title: Evaluation of the CooperVision, Inc. Fanfilcon A and Enfilcon A Daily Wear Contact Lenses When Used for Frequent Replacement for up to One (1) Month of Daily Wear
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FC150625
Record Dates: First submitted 2015-09-16; First posted 2015-09-21 (Estimated); Results first posted 2017-03-08 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- fanfilcon A (test) (Experimental): Subjects will be randomized to wear fanfilcon A lens (test) for one month of daily wear during the study.
  Interventions: Device: fanfilcon A (test)
- enfilcon A (control) (Active Comparator): Subjects will be randomized to wear enfilcon A lens (control) for one month of daily wear during the study.
  Interventions: Device: enfilcon A (control)

INTERVENTIONS:
Device: fanfilcon A (test) — silicone hydrogel lens
  Arms: fanfilcon A (test)
Device: enfilcon A (control) — silicone hydrogel lens
  Arms: enfilcon A (control)

SUMMARY:
This study is a masked, multi-center, daily wear, monthly replacement, bilateral, randomized, lens blocked (subjects remain in the same lens brand throughout the study) concurrent control study enrolling up to 90 subjects with a study duration of approximately three months. Subjects will be randomized into the study contact lenses in a two to one (2:1) ratio of fanfilcon A lens (test) to enfilcon A lens (control).

DETAILED DESCRIPTION:
Subjects will be randomized into the study contact lenses in a two to one (2:1) ratio of fanfilcon A lens (test) to enfilcon A lens (control). This should result in a study population of approximately 60 test subjects and 30 control subjects.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age as of the date of evaluation for the study.
* Have:

  * Read the Informed Consent
  * Been given an explanation of the Informed Consent
  * Indicated understanding of the Informed Consent
  * Signed the Informed Consent document.
* Be willing and able to adhere to the instructions set forth in this protocol and able to keep all specified appointments.
* Be an adapted, current full-time silicone hydrogel or soft contact lens wearer. An adapted full-time wearer is defined as wearing contact lenses at least 5 days per week for at least 8 hours per day for at least one month prior to participation in the study.
* Possess or obtain prior to dispensing, wearable and visually functional (20/40 or better) eyeglasses.
* Be in good general health, based on his/her knowledge.
* Require spectacle lens powers between -0.50 and -8.00 diopters sphere with no more than 1.50 diopter of refractive astigmatism and be willing to wear contact lenses in both eyes.
* Have manifest refraction Snellen visual acuities (VA) equal to or better than20/25 in each eye.
* To be eligible for lens dispensing, the subject must achieve 20/30 VA or better in each eye with the study lens and the investigator must judge the fit as acceptable or optimal.

Exclusion Criteria:

* Wearing lenses in a monovision modality and is unwilling to be fit with distance lenses in both eyes for the duration of the study. Note: Subjects may not wear lenses in a monovision modality at any time during the study as it will interfere with the visual acuity analysis.
* Poor personal hygiene.
* Any active participation in another clinical trial during this trial or within 30 days prior to this study.
* To the best of the subject's knowledge, she is currently pregnant, is lactating or is planning a pregnancy within the next 3 months.
* A member, relative or household member of the investigator or of the investigational office staff.
* Has a known sensitivity to the ingredients used in the Multi-Purpose Disinfection Lens Care System (MPS) approved for use in the study and is unable or unwilling to use the alternate care system.
* Previous refractive surgery; or current or previous orthokeratology treatment.
* Is aphakic or pseudophakic.
* Ocular or systemic disease such as, but not limited to: anterior uveitis or iritis (past or present), glaucoma, Sjögren's syndrome, lupus erythematosus, scleroderma, keratoconus or uncontrolled diabetes.
* The need for topical ocular medications or any systemic medication which might interfere with contact lens wear or require the lenses to be removed during the day.
* The presence of clinically significant (grade 2, 3 or 4) anterior segment abnormalities; or the presence of any inflammations such as iritis; or any infection of the eye, lids, or associated structures.
* A known history of corneal hypoesthesia (reduced corneal sensitivity), corneal ulcer, corneal infiltrates, iritis, bacterial or fungal infections.
* A history of papillary conjunctivitis that has interfered with contact lens wear.
* Slit lamp findings that would contraindicate contact lens wear, including but not limited to:

  * Pathological dry eye or associated dry eye symptoms with decreased tear levels and punctuate staining > Grade 2
  * Pterygium
  * Corneal scars within the visual axis
  * Neovascularization or ghost vessels > 1.0 mm in from the limbus
  * Giant papillary conjunctivitis (GPC) of > Grade 2
  * Anterior uveitis or iritis
  * Seborrheic eczema, seborrheic conjunctivitis or blepharitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2015-09-21 (Actual); Primary Completion 2016-01-27 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric M White, OD, Principal Investigator — Eric White, O.D., Inc.; Peter T Van Hoven, OD, Principal Investigator — Primary Eyecare Group, P.C.; Amanda L Barker, OD, Principal Investigator — Advanced Family Eye Care; Mark E Nakano, OD, Principal Investigator — Mark Nakano, O.D.; Thomas G Quinn, OD, Principal Investigator — Quinn, Foster & Associates; Mary Jo Stiegemeier, OD, Principal Investigator — Western Reserve Vision Care, Inc
Locations (6):
- United States (6):
  - Eric White, O.D., Inc., San Diego, California
  - Mark Nakano, O.D., Torrance, California
  - Advanced Family Eye Care, Denver, North Carolina
  - Quinn, Foster & Associates, Athens, Ohio
  - Western Reserve Vision Care, Inc., Beachwood, Ohio
  - Primary Eyecare Group, P.C., Brentwood, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were randomized to the study lenses based on a 2 to 1 ratio within each investigational site and across the entire study using randomization tables.
Pre-assignment Details: Two (2) subjects were ineligible and were not randomized and exited the study. This left 90 subjects randomized into the test and control products.
Period: Lens Dispensed
Arm/Group | Fanfilcon A (Test) | Enfilcon A (Control)
Started | 60 | 30
Completed | 60 | 30
Not Completed | 0 | 0
Period: Week 1
Arm/Group | Fanfilcon A (Test) | Enfilcon A (Control)
Started | 60 | 30
Completed | 60 | 30
Not Completed | 0 | 0
Period: Week 2
Arm/Group | Fanfilcon A (Test) | Enfilcon A (Control)
Started | 60 | 30
Completed | 59 | 29
Not Completed | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Period: Month 1
Arm/Group | Fanfilcon A (Test) | Enfilcon A (Control)
Started | 59 | 29
Completed | 58 | 29
Not Completed | 1 | 0
Not completed — Lens Discomfort | 1 | 0
Period: Month 2
Arm/Group | Fanfilcon A (Test) | Enfilcon A (Control)
Started | 58 | 29
Completed | 54 | 29
Not Completed | 4 | 0
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Month 3
Arm/Group | Fanfilcon A (Test) | Enfilcon A (Control)
Started | 54 | 29
Completed | 54 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are collected for all completed subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fanfilcon A (Test) | Enfilcon A (Control) | Total
Number analyzed (Participants) | 60 | 30 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.72 (10.320) | 33.67 (10.162) | 34.37 (10.223)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 23 | 72
  Male | 11 | 7 | 18

OUTCOME MEASURES:

1. Primary Outcome: Epithelial Edema - Fanfilcon A Lens (Test)
Description: Epithelial edema is assessed for fanfilcon A lens (test). Grading Scale 0-4, 0=none, 1=trace, 2=mild, 3=moderate, 4=severe
Time Frame: Baseline, Week 1, Week 2, Month 1, Month 2, Month 3
Population: All sites, test subjects' completed eyes. One subject (2 eyes) data was not collected at 2 week visit. Unscheduled visits included one subject visiting between week 2 and 1 month visit and one subject visiting between months 2 and 3.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Groups:
- Baseline; Week 1; Week 2; Month 1; Month 2; Month 3; Unscheduled: fanfilcon A lens (test)
Arm/Group | Baseline | Week 1 | Week 2 | Month 1 | Month 2 | Month 3 | Unscheduled
Number analyzed (Participants) | 54 | 54 | 53 | 54 | 54 | 54 | 2
Number analyzed (Eyes) | 108 | 108 | 106 | 108 | 108 | 108 | 4
percentage of eyes
  None | 100.0 | 100.0 | 99.1 | 100.0 | 100.0 | 100.0 | 100.0
  Trace | 0.0 | 0.0 | 0.9 | 0.0 | 0.0 | 0.0 | 0.0
  Mild | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Moderate | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Severe | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

2. Primary Outcome: Epithelial Edema - Enfilcon A Lens (Control)
Description: Epithelial edema is assessed for enfilcon A lens (control). Grading scale 0-4, 0=none, 1=trace, 2=mild, 3=moderate, 4=severe
Time Frame: Baseline, Week 1, Week 2, Month 1, Month 2, Month 3
Population: All sites, control completed subjects' eyes Three subjects (6 eyes) data were not collected during Week 1 visit. One subject (2 eyes) data was not collected during Month 2 visit. Unscheduled visits included: 2 subjects visiting between weeks 1 and 2, and one subject visiting between months 2 and 3.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Groups:
- Baseline; Week 1; Week 2; Month 1; Month 2; Month 3; Unscheduled: enfilcon A lens (control)
Arm/Group | Baseline | Week 1 | Week 2 | Month 1 | Month 2 | Month 3 | Unscheduled
Number analyzed (Participants) | 29 | 26 | 29 | 29 | 28 | 29 | 3
Number analyzed (Eyes) | 58 | 52 | 58 | 58 | 56 | 58 | 6
percentage of eyes
  None | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0
  Trace | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  MIld | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Moderate | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Severe | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

3. Primary Outcome: Stromal Edema - Fanfilcon A Lens (Test)
Description: Stromal edema is assessed for fanfilcon A lens (test). Grading Scale 0-4, 0=none, 1=trace, 2=mild, 3=moderate, 4=severe
Time Frame: Baseline, Week 1, Week 2, Month 1, Month 2, Month 3
Population: All sites, test subjects' completed eyes. One subject (2 eyes) data was not collected during at 2 week visit. Unscheduled visits included one subject visiting between week 2 and 1 month visit and one subject visiting between months 2 and 3.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Baseline | Week 1 | Week 2 | Month 1 | Month 2 | Month 3 | Unscheduled
Number analyzed (Participants) | 54 | 54 | 53 | 54 | 54 | 54 | 2
Number analyzed (Eyes) | 108 | 108 | 106 | 108 | 108 | 108 | 4
percentage of eyes
  None | 100.0 | 100.0 | 99.1 | 100.0 | 100.0 | 100.0 | 100.0
  Trace | 0.0 | 0.0 | 0.9 | 0.0 | 0.0 | 0.0 | 0.0
  Mild | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Moderate | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Severe | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

4. Primary Outcome: Stromal Edema - Enfilcon A Lens (Control)
Description: Stromal edema is assessed for enfilcon A lens (control). Grading Scale 0-4, 0=none, 1=trace, 2=mild, 3=moderate, 4=severe
Time Frame: Baseline, Week 1, Week 2, Month 1, Month 2, Month 3
Population: as for outcome 2
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Baseline | Week 1 | Week 2 | Month 1 | Month 2 | Month 3 | Unscheduled
Number analyzed (Participants) | 29 | 26 | 29 | 29 | 28 | 29 | 3
Number analyzed (Eyes) | 58 | 52 | 58 | 58 | 56 | 58 | 6
percentage of eyes
  None | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0
  Trace | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Mild | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Moderate | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Severe | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

5. Primary Outcome: Corneal Infiltrates - Fanfilcon A Lens (Test)
Description: Corneal infiltrates is assessed for fanfilcon A lens (test). Grading scale: Absent/present
Time Frame: Baseline, Week 1, Week 2, Month 1, Month 2, Month 3
Population: as for outcome 1
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Baseline | Week 1 | Week 2 | Month 1 | Month 2 | Month 3 | Unscheduled
Number analyzed (Participants) | 54 | 54 | 53 | 54 | 54 | 54 | 2
Number analyzed (Eyes) | 108 | 108 | 106 | 108 | 108 | 108 | 4
percentage of eyes
  Absent | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0
  Present | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

6. Primary Outcome: Corneal Infiltrates - Enfilcon A Lens (Control)
Description: Corneal infiltrates is assessed for enfilcon A lens (control). Grading scale: absent/present
Time Frame: Baseline, Week 1, Week 2, Month 1, Month 2, Month 3
Population: as for outcome 2
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Baseline | Week 1 | Week 2 | Month 1 | Month 2 | Month 3 | Unscheduled
Number analyzed (Participants) | 29 | 26 | 29 | 29 | 28 | 29 | 3
Number analyzed (Eyes) | 58 | 52 | 58 | 58 | 56 | 58 | 6
percentage of eyes
  Absent | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0
  Present | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

7. Primary Outcome: Corneal Vascularization - Fanfilcon A Lens (Test)
Description: Corneal vascularization is assessed for fanfilcon A lens (test). Grading Scale 0-4, 0=none, 1=trace, 2=mild, 3=moderate, 4=severe
Time Frame: Baseline, Week 1, Week 2, Month 1, Month 2, Month 3
Population: as for outcome 1
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Baseline | Week 1 | Week 2 | Month 1 | Month 2 | Month 3 | Unscheduled
Number analyzed (Participants) | 54 | 54 | 53 | 54 | 54 | 54 | 2
Number analyzed (Eyes) | 108 | 108 | 106 | 108 | 108 | 108 | 4
percentage of eyes
  None | 90.7 | 92.6 | 92.5 | 92.6 | 94.4 | 91.7 | 100.0
  Trace | 9.3 | 7.4 | 7.5 | 7.4 | 5.6 | 8.3 | 0.0
  Mild | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Moderate | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Severe | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

8. Primary Outcome: Corneal Vascularization - Enfilcon A Lens (Control)
Description: Corneal vascularization is assessed for enfilcon A lens (control). Grading Scale 0-4, 0=none, 1=trace, 2=mild, 3=moderate, 4=severe
Time Frame: Baseline, Week 1, Week 2, Month 1, Month 2, Month 3
Population: All sites, control completed subjects' eyes. Three subjects (6 eyes) data were not collected during Week 1 visit. One subject (2 eyes) data was not collected during Month 2 visit. Unscheduled visits included: 2 subjects visiting between weeks 1 and 2, and one subject visiting between months 2 and 3.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Baseline | Week 1 | Week 2 | Month 1 | Month 2 | Month 3 | Unscheduled
Number analyzed (Participants) | 29 | 26 | 29 | 29 | 28 | 29 | 3
Number analyzed (Eyes) | 58 | 52 | 58 | 58 | 56 | 58 | 6
percentage of eyes
  None | 86.2 | 92.3 | 93.1 | 93.1 | 96.4 | 96.6 | 100.0
  Trace | 13.8 | 7.7 | 6.9 | 6.9 | 3.6 | 3.4 | 0.0
  Mild | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Moderate | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Severe | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

9. Primary Outcome: Corneal Staining - Fanfilcon A Lens (Test)
Description: Corneal staining with fluorescein is assessed for fanfilcon A lens (test). Grading Scale 0-4, 0=none, 1=trace, 2=mild, 3=moderate, 4=severe; Grading regions: S - Superior, T - Temporal, C - Central, N - Nasal, I - Inferior;
Time Frame: Baseline, Week 1, Week 2, Month 1, Month 2, Month 3
Population: as for outcome 1
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Baseline | Week 1 | Week 2 | Month 1 | Month 2 | Month 3 | Unscheduled
Number analyzed (Participants) | 54 | 54 | 53 | 54 | 54 | 54 | 2
Number analyzed (Eyes) | 108 | 108 | 106 | 108 | 108 | 108 | 4
percentage of eyes
  Superior - None | 96.3 | 92.6 | 93.4 | 93.5 | 97.2 | 96.3 | 100.0
  Superior - Trace | 3.7 | 7.4 | 2.8 | 6.5 | 2.8 | 2.8 | 0.0
  Superior - Mild | 0.0 | 0.0 | 3.8 | 0 | 0 | 0.9 | 0.0
  Superior - Moderate | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Superior - Severe | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Temporal - None | 93.5 | 97.2 | 95.3 | 96.3 | 92.6 | 90.7 | 100.0
  Temporal - Trace | 6.5 | 2.8 | 3.8 | 2.8 | 5.6 | 8.3 | 0.0
  Temporal - Mild | 0.0 | 0.0 | 0.9 | 0.9 | 1.9 | 0.9 | 0.0
  Temporal - Moderate | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Temporal - Severe | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Central - None | 94.4 | 88.9 | 88.7 | 88.0 | 95.4 | 88.9 | 100.0
  Central - Trace | 5.6 | 11.1 | 10.4 | 11.1 | 2.8 | 11.1 | 0.0
  Central - Mild | 0.0 | 0.0 | 0.9 | 0.9 | 1.9 | 0.0 | 0.0
  Central - Moderate | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Central - Severe | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Nasal - None | 90.7 | 90.7 | 96.2 | 92.6 | 95.4 | 96.3 | 100.0
  Nasal - Trace | 9.3 | 7.4 | 3.8 | 5.6 | 3.7 | 3.7 | 0.0
  Nasal - Mild | 0.0 | 1.9 | 0.0 | 1.9 | 0.9 | 0.0 | 0.0
  Nasal - Moderate | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Nasal - Severe | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Inferior - None | 70.4 | 70.4 | 71.7 | 74.1 | 67.6 | 70.4 | 100.0
  Inferior - Trace | 29.6 | 28.7 | 21.7 | 17.6 | 23.1 | 23.1 | 0.0
  Inferior - Mild | 0.0 | 0.9 | 6.6 | 8.3 | 9.3 | 6.5 | 0.0
  Inferior - Moderate | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Inferior - Severe | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

10. Primary Outcome: Corneal Staining - Enfilcon A Lens (Control)
Description: Corneal staining with fluorescein is assessed for enfilcon A lens (control). Grading Scale 0-4, 0=none, 1=trace, 2=mild, 3=moderate, 4=severe; Grading regions: S - Superior, T - Temporal, C - Central, N - Nasal, I - Inferior;
Time Frame: Baseline, Week 1, Week 2, Month 1, Month 2, Month 3
Population: as for outcome 8
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Baseline | Week 1 | Week 2 | Month 1 | Month 2 | Month 3 | Unscheduled
Number analyzed (Participants) | 29 | 26 | 29 | 29 | 28 | 29 | 3
Number analyzed (Eyes) | 58 | 52 | 58 | 58 | 56 | 58 | 6
percentage of eyes
  Superior - None | 75.9 | 84.6 | 96.6 | 93.1 | 78.6 | 93.1 | 100.0
  Superior - Trace | 24.1 | 15.4 | 3.4 | 6.9 | 21.4 | 6.9 | 0.0
  Superior - Mild | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Superior - Moderate | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Superior - Severe | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Temporal - None | 65.5 | 84.6 | 75.9 | 89.7 | 75.0 | 89.6 | 100.0
  Temporal - Trace | 34.5 | 15.4 | 24.1 | 10.3 | 25.0 | 10.3 | 0.0
  Temporal - Mild | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 6.9 | 0.0
  Temporal - Moderate | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Temporal - Severe | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Central - None | 62.1 | 73.1 | 79.3 | 75.8 | 85.7 | 82.8 | 83.4
  Central - Trace | 37.9 | 26.9 | 20.7 | 24.1 | 14.3 | 17.2 | 8.3
  Central - Mild | 0.0 | 0.0 | 0.0 | 3.4 | 0.0 | 0.0 | 8.3
  Central - Moderate | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Central - Severe | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Nasal - None | 62.1 | 73.0 | 65.5 | 79.3 | 78.6 | 75.9 | 100.0
  Nasal - Trace | 37.9 | 26.9 | 34.5 | 20.7 | 21.4 | 24.1 | 0.0
  Nasal - Mild | 0.0 | 3.8 | 0.0 | 0.0 | 0.0 | 1.8 | 0.0
  Nasal - Moderate | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Nasal - Severe | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Inferior - None | 51.7 | 57.6 | 27.6 | 62.0 | 53.5 | 44.8 | 66.7
  Inferior - Trace | 48.3 | 42.3 | 72.4 | 37.9 | 46.4 | 55.2 | 33.3
  Inferior - Mild | 0.0 | 7.7 | 3.4 | 10.3 | 3.6 | 3.4 | 0.0
  Inferior - Moderate | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Inferior - Superior | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

11. Primary Outcome: Limbal Hyperemia - Fanfilcon A Lens (Test)
Description: Limbal hyperemia is assessed for fanfilcon A lens (test). Grading Scale 0-4, 0=none, 1=trace, 2=mild, 3=moderate, 4=severe
Time Frame: Baseline, Week 1, Week 2, Month 1, Month 2, Month 3
Population: as for outcome 1
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Baseline | Week 1 | Week 2 | Month 1 | Month 2 | Month 3 | Unscheduled
Number analyzed (Participants) | 54 | 54 | 53 | 54 | 54 | 54 | 2
Number analyzed (Eyes) | 108 | 108 | 106 | 108 | 108 | 108 | 4
percentage of eyes
  None | 80.6 | 88.9 | 76.4 | 80.6 | 82.4 | 75.9 | 100.0
  Trace | 19.4 | 11.1 | 23.6 | 19.4 | 17.6 | 23.1 | 0.0
  Mild | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.9 | 0.0
  Moderate | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Severe | 0.0 | 0.0 | 0 | 0.0 | 0.0 | 0.0 | 0.0

12. Primary Outcome: Limbal Hyperemia - Enfilcon A Lens (Control)
Description: Limbal hyperemia is assessed for enfilcon A lens (control). Grading Scale 0-4, 0=none, 1=trace, 2=mild, 3=moderate, 4=severe
Time Frame: Baseline, Week 1, Week 2, Month 1, Month 2, Month 3
Population: as for outcome 2
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Baseline | Week 1 | Week 2 | Month 1 | Month 2 | Month 3 | Unscheduled
Number analyzed (Participants) | 29 | 26 | 29 | 29 | 28 | 29 | 3
Number analyzed (Eyes) | 58 | 52 | 58 | 58 | 56 | 58 | 6
percentage of eyes
  None | 79.3 | 80.8 | 93.1 | 93.1 | 92.9 | 87.9 | 100.0
  Trace | 20.7 | 19.2 | 6.9 | 6.9 | 7.1 | 10.3 | 0.0
  Mild | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 1.7 | 0.0
  Moderate | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Severe | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

13. Primary Outcome: Bulbar Hyperemia - Fanfilcon A Lens (Test)
Description: Bulbar hyperemia is assessed for fanfilcon A lens (test). Grading Scale 0-4, 0=none, 1=trace, 2=mild, 3=moderate, 4=severe
Time Frame: Baseline, Week 1, Week 2, Month 1, Month 2, Month 3
Population: as for outcome 1
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Baseline | Week 1 | Week 2 | Month 1 | Month 2 | Month 3 | Unscheduled
Number analyzed (Participants) | 54 | 54 | 53 | 54 | 54 | 54 | 2
Number analyzed (Eyes) | 108 | 108 | 106 | 108 | 108 | 108 | 4
percentage of eyes
  None | 60.2 | 77.8 | 67.0 | 68.5 | 73.1 | 69.4 | 66.7
  Trace | 39.8 | 21.3 | 32.1 | 31.5 | 26.9 | 29.6 | 33.3
  Mild | 0.0 | 0.9 | 0.9 | 0.0 | 0.0 | 0.9 | 0.0
  Moderate | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Severe | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

14. Primary Outcome: Bulbar Hyperemia - Enfilcon A Lens (Control)
Description: Bulbar hyperemia is assessed for enfilcon A lens (control). Grading Scale 0-4, 0=none, 1=trace, 2=mild, 3=moderate, 4=severe
Time Frame: Baseline, Week 1, Week 2, Month 1, Month 2, Month 3
Population: as for outcome 8
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Baseline | Week 1 | Week 2 | Month 1 | Month 2 | Month 3 | Unscheduled
Number analyzed (Participants) | 29 | 26 | 29 | 29 | 28 | 29 | 3
Number analyzed (Eyes) | 58 | 52 | 58 | 58 | 56 | 58 | 6
percentage of eyes
  None | 65.5 | 61.5 | 72.4 | 69.0 | 92.9 | 81.0 | 100.0
  Trace | 34.5 | 38.5 | 27.6 | 31.0 | 7.1 | 17.2 | 0.0
  Mild | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 1.7 | 0.0
  Moderate | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Severe | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

15. Primary Outcome: Palpebral Conjunctiva - Fanfilcon A Lens (Test)
Description: Palpebral conjunctiva is assessed for fanfilcon A lens (test). Grading scale: Absent/present
Time Frame: Baseline, Week 1, Week 2, Month 1, Month 2, Month 3
Population: as for outcome 1
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Baseline | Week 1 | Week 2 | Month 1 | Month 2 | Month 3 | Unscheduled
Number analyzed (Participants) | 54 | 54 | 53 | 54 | 54 | 54 | 2
Number analyzed (Eyes) | 108 | 108 | 106 | 108 | 108 | 108 | 4
percentage of eyes
  Absent | 69.4 | 64.8 | 63.2 | 67.6 | 60.2 | 58.3 | 50.0
  Present | 30.6 | 35.2 | 36.8 | 32.4 | 39.8 | 41.7 | 50.0

16. Primary Outcome: Palpebral Conjunctiva - Enfilcon A Lens (Control)
Description: Palpebral conjunctiva is assessed for enfilcon A lens (control). Grading scale: absent/present
Time Frame: Baseline, Week 1, Week 2, Month 1, Month 2, Month 3
Population: as for outcome 8
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Baseline | Week 1 | Week 2 | Month 1 | Month 2 | Month 3 | Unscheduled
Number analyzed (Participants) | 29 | 26 | 29 | 29 | 28 | 29 | 3
Number analyzed (Eyes) | 58 | 52 | 58 | 58 | 56 | 58 | 6
percentage of eyes
  Absent | 55.2 | 69.2 | 62.1 | 58.6 | 67.9 | 67.2 | 66.7
  Present | 44.8 | 30.8 | 37.9 | 41.4 | 32.1 | 32.8 | 33.3

17. Primary Outcome: Visual Acuity - Fanfilcon A Lens (Test)
Description: Visual acuity is assessed for fanfilcon A lens (test) using Snellen chart.
Time Frame: Week 1, Week 2, Month 1, Month 2, Month 3
Population: All sites, test subjects' completed eyes. One subject (2 eyes) data was not collected at 2 week visit.
Measure: Number; unit: eyes
Units Other Than Participants: Eyes
Arm/Group | Week 1 | Week 2 | Month 1 | Month 2 | Month 3
Number analyzed (Participants) | 54 | 53 | 54 | 54 | 54
Number analyzed (Eyes) | 108 | 106 | 108 | 108 | 108
eyes
  20/15 | 27 | 26 | 27 | 27 | 27
  20/20 | 78 | 77 | 78 | 78 | 78
  20/25 | 3 | 3 | 3 | 3 | 3
  20/30 | 0 | 0 | 0 | 0 | 0
  20/40 | 0 | 0 | 0 | 0 | 0
  20/50 | 0 | 0 | 0 | 0 | 0
  20/60 | 0 | 0 | 0 | 0 | 0

18. Primary Outcome: Visual Acuity - Enfilcon A Lens (Control)
Description: Visual acuity is assessed for enfilcon A lens (control) using Snellen chart.
Time Frame: Week 1, Week 2, Month 1, Month 2, Month 3
Population: All sites, control completed subjects' eyes. Three subjects (6 eyes) data were not collected during Week 1 visit. One subject (2 eyes) data was not collected during Month 2 visit.
Measure: Number; unit: eyes
Units Other Than Participants: Eyes
Arm/Group | Week 1 | Week 2 | Month 1 | Month 2 | Month 3
Number analyzed (Participants) | 26 | 29 | 29 | 28 | 29
Number analyzed (Eyes) | 52 | 58 | 58 | 56 | 58
eyes
  20/15 | 14 | 14 | 14 | 14 | 14
  20/20 | 36 | 42 | 42 | 40 | 42
  20/25 | 2 | 2 | 2 | 2 | 2
  20/30 | 0 | 0 | 0 | 0 | 0
  20/40 | 0 | 0 | 0 | 0 | 0
  20/50 | 0 | 0 | 0 | 0 | 0
  20/60 | 0 | 0 | 0 | 0 | 0

19. Primary Outcome: Average Wearing Time - Fanfilcon A Lens (Test)
Description: Average lens wearing time for fanfilcon A lens (test) measured in hours.
Time Frame: Baseline, Week 1, Week 2, Month 1, Month 2, Month 3
Population: All sites, test subjects' completed eyes. One subject data was not collected at 2 week visit. Unscheduled visits included one subject visiting between week 2 and 1 month visit and one subject visiting between months 2 and 3.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Baseline | Week 1 | Week 2 | Month 1 | Month 2 | Month 3 | Unscheduled
Number analyzed (Participants) | 54 | 54 | 53 | 54 | 54 | 54 | 2
hours | 14.17 (4.24) | 13.25 (2.56) | 13.08 (2.23) | 13.18 (2.59) | 13.21 (2.41) | 13.13 (2.61) | 16.50 (0.71)

20. Primary Outcome: Average Wearing Time - Enfilcon A Lens (Control)
Description: Average lens wearing time for enfilcon A lens (control) measured in hours.
Time Frame: Baseline, Week 1, Week 2, Month 1, Month 2, Month 3
Population: All sites, control completed subjects' eyes. Three subjects data was not collected during Week 1 visit. One subject data was not collected during Month 2 visit. Unscheduled visits included: 2 subjects visiting between weeks 1 and 2, and one subject visiting between months 2 and 3.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Baseline | Week 1 | Week 2 | Month 1 | Month 2 | Month 3 | Unscheduled
Number analyzed (Participants) | 29 | 26 | 29 | 29 | 28 | 29 | 3
hours | 13.81 (2.95) | 13.67 (2.58) | 13.41 (2.28) | 13.52 (2.11) | 13.20 (2.50) | 13.62 (2.35) | 12.67 (1.16)

21. Secondary Outcome: Comfort - Fanfilcon A Lens (Test)
Description: Fanfilcon A lens (test) are assessed regarding comfort for the following: comfort upon insertion (CUI), comfort during the day (CDD), end of the day comfort (EDC), overall comfort (OC), and comfort at visit (CV). Subjects were asked to rate comfort from 0-5 (0=excellent, 1=very comfortable, 2=comfortable, 3=slightly uncomfortable, 4=very uncomfortable, or 5=causes pain).
Time Frame: Baseline, Week 1, Week 2, Month 1, Month 2, Month 3
Population: as for outcome 19
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Baseline | Week 1 | Week 2 | Month 1 | Month 2 | Month 3 | Unscheduled
Number analyzed (Participants) | 54 | 54 | 53 | 54 | 54 | 54 | 2
Number analyzed (Eyes) | 108 | 108 | 106 | 108 | 108 | 108 | 4
Eyes
  CUI - excellent | 50 | 50 | 67 | 61 | 60 | 64 | 4
  CUI - very comfortable | 40 | 50 | 29 | 36 | 40 | 40 | 0
  CUI - comfortable | 15 | 6 | 6 | 10 | 6 | 2 | 0
  CUI- slightly uncomfortable | 3 | 2 | 4 | 1 | 2 | 2 | 0
  CUI - very uncomfortable | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CUI - causes pain | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CDD - excellent | 45 | 45 | 48 | 50 | 48 | 48 | 2
  CDD - very comfortable | 38 | 50 | 47 | 40 | 48 | 50 | 2
  CDD - comfortable | 19 | 13 | 9 | 9 | 8 | 6 | 0
  CDD - slightly uncomfortable | 6 | 0 | 0 | 9 | 4 | 4 | 0
  CDD-very uncomfortable | 0 | 0 | 2 | 0 | 0 | 0 | 0
  CDD - causes pain | 0 | 0 | 0 | 0 | 0 | 0 | 0
  EDC - excellent | 14 | 32 | 31 | 30 | 36 | 30 | 2
  EDC - very comfortable | 46 | 34 | 43 | 38 | 32 | 44 | 2
  EDC - comfortable | 27 | 32 | 30 | 22 | 25 | 24 | 0
  EDC - slightly uncomfortable | 19 | 8 | 2 | 16 | 11 | 8 | 0
  EDC - very uncomfortable | 2 | 2 | 0 | 2 | 4 | 2 | 0
  EDC - causes pain | 0 | 0 | 0 | 0 | 0 | 0 | 0
  OC - excellent | 37 | 40 | 40 | 43 | 46 | 46 | 2
  OC - very comfortable | 47 | 58 | 54 | 44 | 42 | 48 | 2
  OC - comfortable | 20 | 8 | 10 | 14 | 14 | 8 | 0
  OC - slightly uncomfortable | 4 | 2 | 0 | 7 | 6 | 6 | 0
  OC - very uncomfortable | 0 | 0 | 2 | 0 | 0 | 0 | 0
  OC - causes pain | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CV - excellent | 60 | 60 | 63 | 56 | 56 | 62 | 2
  CV - very comfortable | 22 | 36 | 30 | 38 | 36 | 34 | 2
  CV - comfortable | 17 | 12 | 11 | 6 | 12 | 8 | 0
  CV - slightly uncomfortable | 7 | 0 | 0 | 6 | 4 | 4 | 0
  CV - very uncomfortable | 2 | 0 | 2 | 2 | 0 | 0 | 0
  CV - causes pain | 0 | 0 | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Comfort - Enfilcon A Lens (Control)
Description: Enfilcon A lens (control) are assessed regarding comfort for the following: comfort upon insertion (CUI), comfort during the day (CDD), end of the day comfort (EDC), overall comfort (OC), and comfort at visit (CV). Subjects were asked to rate comfort from 0-5 (0=excellent, 1=very comfortable, 2=comfortable, 3=slightly uncomfortable, 4=very uncomfortable, or 5=causes pain).
Time Frame: Baseline, 1 week, 2 weeks, 1 month, 2 months, 3 months follow-up
Population: All sites, control completed subjects. Three subjects data was not collected during Week 1 visit. One subject data was not collected during Month 2 visit.
  Unscheduled visits included: 2 subjects visiting between weeks 1 and 2, and one subject visiting between months 2 and 3.
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Baseline | Week 1 | Week 2 | Month 1 | Month 2 | Month 3 | Unscheduled
Number analyzed (Participants) | 29 | 26 | 29 | 29 | 28 | 29 | 3
Number analyzed (eyes) | 58 | 52 | 58 | 58 | 56 | 58 | 6
eyes
  CUI - excellent | 20 | 16 | 30 | 20 | 28 | 26 | 6
  CUI - very comfortable | 26 | 23 | 16 | 24 | 12 | 18 | 0
  CUI - comfortable | 6 | 6 | 12 | 11 | 12 | 12 | 0
  CUI- slightly uncomfortable | 6 | 7 | 0 | 3 | 4 | 2 | 0
  CUI - very uncomfortable | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CUI - causes pain | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CDD - excellent | 26 | 22 | 24 | 18 | 22 | 19 | 6
  CDD - very comfortable | 18 | 15 | 13 | 10 | 17 | 18 | 0
  CDD - comfortable | 12 | 12 | 19 | 20 | 13 | 10 | 0
  CDD - slightly uncomfortable | 2 | 3 | 2 | 10 | 4 | 9 | 0
  CDD-very uncomfortable | 0 | 0 | 0 | 0 | 0 | 2 | 0
  CDD - causes pain | 0 | 0 | 0 | 0 | 0 | 0 | 0
  EDC - excellent | 16 | 12 | 22 | 14 | 16 | 14 | 6
  EDC - very comfortable | 12 | 14 | 5 | 8 | 15 | 12 | 0
  EDC - comfortable | 14 | 10 | 24 | 20 | 15 | 10 | 0
  EDC - slightly uncomfortable | 10 | 14 | 7 | 12 | 8 | 19 | 0
  EDC - very uncomfortable | 6 | 2 | 0 | 4 | 2 | 3 | 0
  EDC - causes pain | 0 | 0 | 0 | 0 | 0 | 0 | 0
  OC - excellent | 20 | 16 | 20 | 18 | 24 | 18 | 4
  OC - very comfortable | 24 | 16 | 19 | 12 | 12 | 16 | 2
  OC- comfortable | 10 | 10 | 16 | 22 | 14 | 16 | 0
  OC - slightly uncomfortable | 4 | 10 | 3 | 6 | 6 | 6 | 0
  OC - very uncomfortable | 0 | 0 | 0 | 0 | 0 | 2 | 0
  OC - causes pain | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CV - excellent | 22 | 28 | 32 | 26 | 32 | 22 | 4
  CV - very comfortable | 16 | 14 | 8 | 16 | 8 | 22 | 0
  CV - comfortable | 12 | 8 | 16 | 14 | 12 | 11 | 2
  CV - slightly uncomfortable | 8 | 2 | 2 | 2 | 4 | 3 | 0
  CV - very uncomfortable | 0 | 0 | 0 | 0 | 0 | 0 | 0
  CV - causes pain | 0 | 0 | 0 | 0 | 0 | 0 | 0

23. Secondary Outcome: Overall Vision Quality - Fanfilcon A Lens (Test)
Description: Overall vision quality (OVQ) and vision at night (VAN) is assessed at the specific time points. Subjects were asked to rate vision from 0-5, (0=excellent, 1=very good, 2=good, 3=poor, 4=very poor, 5= unacceptable).
Time Frame: Baseline, Week 1, Week 2, Month 1, Month 2, Month 3
Population: All sites, test subjects' completed. One subject data was not collected at 2 week visit.
  Unscheduled visits included one subject visiting between week 2 and 1 month visit and one subject visiting between months 2 and 3.
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Baseline | Week 1 | Week 2 | Month 1 | Month 2 | Month 3 | Unscheduled
Number analyzed (Participants) | 54 | 54 | 53 | 54 | 54 | 54 | 2
Number analyzed (eyes) | 108 | 108 | 106 | 108 | 108 | 108 | 4
eyes
  OVC - excellent | 53 | 70 | 68 | 64 | 64 | 70 | 4
  OVC - very good | 41 | 30 | 27 | 28 | 30 | 32 | 0
  OVC - good | 8 | 8 | 9 | 16 | 11 | 4 | 0
  OVC - poor | 6 | 0 | 0 | 0 | 2 | 2 | 0
  OVC - very poor | 0 | 0 | 2 | 0 | 0 | 0 | 0
  OVC - unacceptable | 0 | 0 | 0 | 0 | 1 | 0 | 0
  VAN - excellent | 41 | 60 | 58 | 50 | 52 | 60 | 4
  VAN - very good | 33 | 34 | 32 | 32 | 34 | 32 | 0
  VAN - good | 28 | 14 | 14 | 26 | 22 | 12 | 0
  VAN - poor | 4 | 0 | 2 | 0 | 0 | 4 | 0
  VAN - very poor | 0 | 0 | 0 | 0 | 0 | 0 | 0
  VAN - unacceptable | 2 | 0 | 0 | 0 | 0 | 0 | 0

24. Secondary Outcome: Overall Vision Quality - Enfilcon A Lens (Control)
Description: as for outcome 23
Time Frame: Baseline, Week 1, Week 2, Month 1, Month 2, Month 3
Population: as for outcome 22
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Baseline | Week 1 | Week 2 | Month 1 | Month 2 | Month 3 | Unscheduled
Number analyzed (Participants) | 29 | 26 | 29 | 29 | 28 | 29 | 3
Number analyzed (eyes) | 58 | 52 | 58 | 58 | 56 | 58 | 6
eyes
  OVC - excellent | 23 | 28 | 28 | 22 | 30 | 25 | 4
  OVC - very good | 24 | 10 | 17 | 20 | 15 | 16 | 0
  OVC - good | 11 | 12 | 12 | 14 | 9 | 12 | 2
  OVC - poor | 0 | 2 | 1 | 2 | 0 | 4 | 0
  OVC - very poor | 0 | 0 | 0 | 0 | 2 | 1 | 0
  OVC - unacceptable | 0 | 0 | 0 | 0 | 0 | 0 | 0
  VAN - excellent | 13 | 26 | 28 | 22 | 20 | 20 | 4
  VAN - very good | 26 | 12 | 15 | 18 | 21 | 16 | 2
  VAN - good | 19 | 12 | 14 | 14 | 11 | 18 | 0
  VAN - poor | 0 | 2 | 1 | 4 | 2 | 4 | 0
  VAN - very poor | 0 | 0 | 0 | 0 | 2 | 0 | 0
  VAN- unacceptable | 0 | 0 | 0 | 0 | 0 | 0 | 0

25. Secondary Outcome: Ease of Insertion and Removal - Fanfilcon A Lens (Test)
Description: Ease of Insertion (EOI) and removal (EOR) was assessed. Subjects were asked to rate ease of insertion and removal on scale 0-5 (0=excellent, 1=very good, 2=good, 3=poor, 4=very poor, or 5=unmanageable.
Time Frame: Baseline, Week 1, Week 2, Month 1, Month 2, Month 3
Population: as for outcome 19
Measure: Count of Units; unit: eyes
Units Other Than Participants: eyes
Arm/Group | Baseline | Week 1 | Week 2 | Month 1 | Month 2 | Month 3 | Unscheduled
Number analyzed (Participants) | 54 | 54 | 53 | 54 | 54 | 54 | 2
Number analyzed (eyes) | 108 | 108 | 106 | 108 | 108 | 108 | 4
eyes
  EOI - excellent | 78 | 70 | 72 | 73 | 68 | 72 | 2
  EOI - very good | 26 | 34 | 30 | 30 | 34 | 32 | 2
  EOI - good | 4 | 4 | 2 | 2 | 6 | 4 | 0
  EOI - poor | 0 | 0 | 0 | 3 | 0 | 0 | 0
  EOI - very poor | 0 | 0 | 2 | 0 | 0 | 0 | 0
  EOI - unmanageable | 0 | 0 | 0 | 0 | 0 | 0 | 0
  EOR - excellent | 72 | 62 | 57 | 48 | 58 | 56 | 2
  EOR - very good | 28 | 31 | 33 | 43 | 30 | 30 | 2
  EOR - good | 8 | 11 | 12 | 15 | 18 | 22 | 0
  EOR - poor | 0 | 4 | 2 | 2 | 2 | 0 | 0
  EOR - very poor | 0 | 0 | 2 | 0 | 0 | 0 | 0
  EOR - unmanageable | 0 | 0 | 0 | 0 | 0 | 0 | 0

26. Secondary Outcome: Ease of Insertion and Removal - Enfilcon A Lens (Control)
Description: as for outcome 25
Time Frame: Baseline, Week 1, Week 2, Month 1, Month 2, Month 3
Population: as for outcome 20
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Groups:
- Unscheduled: Unscheduled visits included: 2 subjects visiting between weeks 1 and 2, and one subject visiting between months 2 and 3.
Arm/Group | Baseline | Week 1 | Week 2 | Month 1 | Month 2 | Month 3 | Unscheduled
Number analyzed (Participants) | 29 | 26 | 29 | 29 | 28 | 29 | 3
Number analyzed (Eyes) | 58 | 52 | 58 | 58 | 56 | 58 | 6
Eyes
  EOI - excellent | 34 | 31 | 36 | 30 | 36 | 30 | 6
  EOI - very good | 12 | 14 | 12 | 16 | 10 | 17 | 0
  EOI - good | 10 | 5 | 10 | 10 | 6 | 7 | 0
  EOI - poor | 2 | 2 | 0 | 2 | 4 | 4 | 0
  EOI - very poor | 0 | 0 | 0 | 0 | 0 | 0 | 0
  EOI - unmanageable | 0 | 0 | 0 | 0 | 0 | 0 | 0
  EOR - excellent | 40 | 36 | 40 | 34 | 36 | 34 | 6
  EOR - very good | 12 | 12 | 12 | 16 | 16 | 14 | 0
  EOR - good | 6 | 2 | 5 | 8 | 4 | 10 | 0
  EOR - poor | 0 | 1 | 1 | 0 | 0 | 0 | 0
  EOR - very poor | 0 | 0 | 0 | 0 | 0 | 0 | 0
  EOR - unmanageable | 0 | 1 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Fanfilcon A (Test) | Enfilcon A (Control)
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/30
Other Adverse Events (participants affected / at risk) | 0/60 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other